CLINICAL TRIAL: NCT02179567
Title: First Line Treatment of Elderly Patients With Advanced or Metastatic NSCLC With Docetaxel and Bevacizumab
Brief Title: Docetaxel Plus Bevacizumab for Elderly Patients With Stage IV NSCLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to poor accrual
Sponsor: Hellenic Oncology Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/10.03
Record Dates: First submitted 2014-06-30; First posted 2014-07-02 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: NSCLC
Keywords: Metastatic NSCLC; Elderly; 1st Line; Bevacizumab-based treatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Doc/Bev (Experimental): Docetaxel/Bevacizumab
  Interventions: Drug: Docetaxel; Drug: Bevacizumab

INTERVENTIONS:
Drug: Docetaxel — Docetaxel: 60mg/m2 i.v on day 1. Cycle repeated ever 3 weeks
Drug: Bevacizumab — Bevacizumab: 7.5 mg/kg, iv on day 1. Cycle repeated every 3 weeks

SUMMARY:
The investigators propose to study the efficacy and safety of the combination of Docetaxel plus Bevacizumab in a Phase II trial of elderly subjects with non-small cell lung cancer

DETAILED DESCRIPTION:
About 50% of newly diagnosed cases of NSCLC concern patients older than 65 years, while 30-40% of cases are diagnosed in patients older than 70 years. Furthermore, recent data suggest that during the last decade, the incidence and mortality of NSCLC has decreased in younger patients, while it has increased among older patients. Based on these observations, it becomes clear that NSCLC represents a significant health problem in elderly patients. However, elderly patients are frequently underrepresented in clinical trials evaluating new treatments in NSCLC. Indeed, more than 75% of patients older than 65 years with metastatic NSCLC never receive any kind of chemotherapy in the daily clinical practice.

According to retrospective data,the addition of bevacizumab to a standard, platinum-based chemotherapy regimen improves overall survival in patients with advanced non-squamous-cell, non-small-cell lung cancer and a good ECOG performance status. In addition, bevacizumab prolongs progression-free survival and improves response rate.

In elderly patients there is a complete lack of prospective data regarding the role of bevacizumab. It is not clear whether elderly patients gain any survival benefit or not and if the addition of bevacizumab to standard chemotherapeutic regimens results in a significant increase in toxicity.

There is a clear need to prospectively evaluate the tolerability of bevacizumab when added to standard first-line chemotherapy of elderly NSCLC patients. Therefore, the investigators propose to study the efficacy in elderly (>70 years) patients treated with cytotoxic chemotherapy in combination with bevacizumab in the context of 1st line treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥70 years old
* Cytologically or histologically documented NSCLC
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (at least one measurable lesion)
* World Health Organisation (WHO) performance status 0-2
* Non-frail patients according to Comprehensive Geriatric Assessment
* No prior chemotherapy
* Life expectancy of at least 12 weeks
* Serum bilirubin less than 1.5 times the upper normal limit
* Aspartate Aminotransferase and Alanine Aminotransferase less than 2.5 times the upper normal limit in the absence of demonstrable liver metastases, or less than 5 times the upper normal limit in the presence of liver metastases
* Serum creatinine less than 1.5 times the upper normal limit and Creatinine Clearance >60 ml/min
* Neutrophil count more than 1.5x 109 /L
* Platelet count more than 100x 109 /L
* Before patient enrollment, written informed consent must be given according to Good Clinical Practice guidelines and national/local regulations.

Exclusion Criteria:

* Hemoptysis
* Central nervous system metastases
* Hemorrhagic diathesis or coagulopathy
* Anticoagulation therapy; regular use of aspirin (>325 mg/d), nonsteroidal anti-inflammatory agents, or other agents known to inhibit platelet function
* Major surgery within 28 days before enrolment
* Clinically significant cardiovascular disease
* Medically uncontrolled hypertension
* Radiological evidence of tumors invading or abutting major blood vessels
* Other co-existing malignancies or malignancies diagnosed within the last 5 years (with the exception of basal cell carcinoma or cervical cancer in situ)
* Any evidence of severe uncontrolled concomitant disease (in the opinion of the investigator)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Disease evaluation at Week 9

SECONDARY OUTCOMES:
Disease control rate | Disease evaluation at Week 9
  Disease control rate is defined as the proportion of patients with complete response or partial response or stable disease for at least 16 weeks
Progression Free Survival | 1 year
Overall Survival | 1 year
Safety Profile | Every three weeks up to 18 weeks
  Patients will be evaluated for Adverse Events (related or unrelated to the treatment) on Day 1 of each cycle (cycle repeated every 3 weeks) up to 18 weeks from the date of first dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Lambros Vamvakas, MD, Principal Investigator — University Hospital of Herklion; Athanasios Karambeazis, MD, Principal Investigator — Medical Oncology Unit NIMTS (Veterans Hospital)
Locations (5):
- Greece (5):
  - University Hospital of Crete, Dep of Medical Oncology Heraklion, Greece, Heraklion, Crete
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - 401 Military Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens Athens, Greece, Athens
  - Medical Oncology Unit NIMTS (Veterans Hospital), Athens